CLINICAL TRIAL: NCT02801110
Title: Comparison of [18F] FDOPA PET/MR Imaging in Patients With Short and Long Standing Parkinson's Disease: Pilot Study
Brief Title: PET/MR Imaging in Patients With Short and Long Standing Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: david groshar (Other)
Responsible Party: Sponsor-Investigator, david groshar, Prof. David Groshar, Assuta Medical Center
Organization: Assuta Medical Center (Other)
Other Study IDs: 0015-16-ASMC
Record Dates: First submitted 2016-06-13; First posted 2016-06-15 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Parkinson's disease (PD) is a chronic, progressive, neurodegenerative disease that affects 1% of the population older than 60 years. The disease presents as a movement disorder manifesting mainly with resting tremor, bradykinesia, cogwheel rigidity and postural instability along with cognitive and behavioral disturbances and symptoms of other non-motor systems dysfunction. The pathophysiology of the motor dysfunction in PD is related to gradual loss of nigrostriatal dopaminergic neurons (originating from the substantia nigra (SN) compacta to the striatum) leading eventually to depletion of dopamine in the striatum.

Striatal fluorine-18 isotopologue for L-3,4-dihydroxyphenylalanine([18F] F-DOPA) uptake follows a typical spatiotemporal pattern along the course of disease starting with a decreased uptake in the dorso-caudal putamen (contralateral to the side of predominant motor involvement) that progress to the caudate nucleus.

The role of traditional magnetic resonance imaging (MRI) in the evaluation of PD is aimed mainly to differentiate idiopathic PD from secondary parkinsonism (e.g. vascular) and from other degenerative but atypical parkinsonian syndromes (e.g.Progressive supranuclear palsy ( PSP), Multiple system atrophy (MSA) etc.) that are associated with distinct structural features and therefore help establishing the diagnosis. However, new MR sequences such as diffuse tensor imaging (DTI) and susceptibility-weighted imaging (SWI) are now being investigated to evaluate the nigrostriatal dopaminergic neurons and iron accumulation in the SN, respectively.

Resting-state functional magnetic resonance imaging (fMRI) that depicts brain network organization has been shown to be altered in patients with PD. In this technique, temporally synchronous, spatially distributed, spontaneous low frequency blood-oxygen level-dependent signal fluctuations in task-free settings are further clustered into maps of functional large-scale neural networks. Lower network efficiency that worsens as disease progresses has been shown in patients with PD.

Recently, it has been shown that the integration of MRI and PET is technically feasible. The investigators believe that PET/MRI offers true multimodality imaging by combining anatomy, function and molecular processes that will allow more accurate identification of disease progression.

To the best of our knowledge, this will be the first study to evaluate idiopathic PD (IPD) with 18F FDOPA PET/MRI.

The aim of the study is to assess the feasibility of the modality and to evaluate both visually and quantitatively the association between the dopamine metabolism measured in the striatum by 18F-FDOPA PET with structural and functional MR findings in patients diagnosed with IPD with asymmetrical motor signs.

DETAILED DESCRIPTION:
Study Objectives and Purpose:

1. To assess the feasibility of 18F FDOPA PET/MR in the setting of IPD.
2. To correlate and compare pattern of dynamic and/or static 18F-FDOPA uptake in the striatum with MR findings.
3. To compare the different variables between the contra and ipsilateral hemispheric side of predominant motor involvement in patients with asymmetric motor disturbances.

Materials and Methods:

Study Design: This is a prospective, pilot, cohort

Study population:

Patients diagnosed with IPD suffering from asymmetrical motor signs.

Participant recruitment:

Eligible consecutive patients, satisfying the inclusion criteria, will be identified and recruited by neurological clinics.

Informed consent: Before enrollment, written informed consent will be obtained from each patient.

Participant Sampling: All patients fulfilling inclusion criteria and providing informed consent will be consecutively enrolled.

Imaging diagnostic PET/MR protocol All scans will be performed in the department of Nuclear Medicine at Tel-Aviv Assuta Medical Center using a PET/MR scanner (Biograph mMR, Siemens AG, Erlangen, Germany) in accordance with the manufacturer's guidelines.

Patients are required to fast at least 4 hours prior to arrival to the department. Upon arrival an intravenous catheter will be placed for radiopharmaceutical and gadolinium administration. Patients will receive an intravenous injection of 10 Millicurie (mCi) of 18F-FDOPA on the PET MR table and scanning will begin immediately. Dynamic PET parameters will be acquired along with the different MR sequences. MR of the brain will include the following sequences: T1, T2 and T2 fluid attenuated inversion recovery sequence (FLAIR), susceptibility-weighted sequences (SWI), blood-oxygenation level-dependent (BOLD) signals for resting-state functional imaging. In addition, perfusion of the brain will be evaluated with and without gadolinium.

For contrast-enhanced sequences the investigators use Dotarem (gadoteric acid)(0.2 ml/kg ,0.1 mmol/kg at 2ml/s, 20ml saline flush) The total scan time will be about 45 minutes.

Data collection:

For eligible patients, the following data will be recorded at baseline.

1. Baseline parameters: date of birth, sex, age at diagnosis and (motor) symptoms onset.
2. Detailed medical history.
3. Physical examination.
4. List of medications (and doses for anti PD and psychiatric medications)
5. Hoehn and Yahr stage.
6. Evaluation using the Movement Disorders Society - performed by neurologist.

MR findings:

* Abnormal structural findings of the brain.
* DTI measurements in the nigrostriatal dopaminergic neuron tracts.
* Iron overload in the SN.
* Comparison of resting-state brain networks in patients with asymmetrical motor signs with normal maps

PET findings:

1. Visual assessment and quantitative measurements of static F-DOPA (e.g.,Standardized Uptake Values (SUV) SUVmax and SUVmean) will be performed in the putamen and caudate nucleus bilaterally.
2. Measurements of dynamic F-DOPA parameters when available ( e.g., time to peak, peak value etc.) will be measured.

Statistics Patient characteristics will be summarized using descriptive statistics. Quantitative variables will be presented as mean and SD, qualitative variables will be presented as frequencies.

Pearson correlation coefficient will be used to measure the strength of the relationship between the PET and the MR parameters.

A t-test will be used to compare the mean values of the different parameters. Sample size: This is a pilot study for which a sample size of 40 patients is required.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 30 below 80 years of age.
2. A clinical diagnosis of idiopathic PD.
3. Patients with asymmetric presentation of PD (by history/medical documentation).
4. Patients with persistent motor asymmetry (with side predominance respecting the side of symptom onset).

Exclusion Criteria:

1. Patients with history of other brain disorder/pathology.
2. Patients with atypical signs suggesting another neurodegenerative disorder, psychiatric disorders, signs of severe cognitive deterioration, severe cardiovascular comorbidity
3. Patients treated with levodopa.
4. Patients on medication known to interfere with the DAT or catechol O-methyltransferase inhibitors, or with dopamine receptor blocking / or catecholamine re-uptake blocking properties.
5. Patients suffering from dystonia.
6. Pregnancy/ Breastfeeding.
7. Contraindication to MR imaging.
8. Uncontrolled head/body movements.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IPD suffering from asymmetrical motor signs.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
correlation between SUV to DTI measurements | 24 months
  non interventional study.

CONTACTS AND LOCATIONS:
Overall Officials: David Groshar, MD, Principal Investigator — Head of nuclear medicine unit in Assuta Medical Centers

IPD SHARING:
Plan to Share IPD: No